CLINICAL TRIAL: NCT00522171
Title: A Randomized, Prospective, Parallel Group Study Comparing the Harmonic™ to Electro Surgery in Lower Body Lift Procedures
Brief Title: Harmonic Versus Electro Surgery in Lower Body Lift Procedures
Acronym: LBL
Status: Terminated | Type: Observational
Why Stopped: This study was terminated early due to lack of adequate enrollment.
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Denise Breiner, Ethicon Endo-Surgery
Other Study IDs: CI-06-0009
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-11

CONDITIONS: Obesity
Keywords: Harmonic; Massive Weight Loss; Electro Surgery; Skin and Fat Redundancy after massive weight loss; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Electro Surgery: Electro Surgical instruments are used to cut and coagulate tissue using alternating electric current at the surgical site. In Electro Surgery, the patient is included in the circuit and current enters the patient's body.
  Interventions: Device: The Harmonic™ ultrasonic scalpel

INTERVENTIONS:
Device: The Harmonic™ ultrasonic scalpel — A surgical instrument that uses ultrasonic energy that allows both cutting and coagulating at the precise point of application.
  Other Names: Harmonic Technology; Manufacturer: Ethicon Endo-Surgery, Inc., Cincinnati, OH.

SUMMARY:
The objective of this study is to determine if the use of The Harmonic™ (an ultrasonic surgical instrument) in Lower Body Lift procedures reduces volume and duration of wound drainage after surgery when compared to Electro Surgery.

DETAILED DESCRIPTION:
Lower Body Lift procedures are performed to correct skin redundancy and muscle diastases caused by significant weight loss, poor skin tone, etc. Lower Body Lift procedures involve a high risk of early complications, including hematomas, seromas, necrosis, and wound-healing problems. The occurrence of these complications may be due in part to the extensive undermining and division of the superficial and the deep arterial systems, done in conventional procedures.

Persistent serous wound drainage and seromas are the most common complications in Lower Body Lift procedures. The rate of serous fluid collection determines the time drains need to remain in place. Although suction drains reduce seroma formation, prolonged use can delay healing, cause injury, and increase the risk of retrograde infection and patient discomfort. Wound drainage has a direct correlation with seroma formation. The loss of protein nutrients and minerals in the serum drained is also a concern with prolonged drainage that can result in healing delays.

The Harmonic™ technology uses ultrasonic energy that allows both cutting and coagulating at the precise point of application. The Harmonic™ has been used since 1992 predominantly in urology and gastro-intestinal surgery (laparoscopic surgery). Significantly reduced serous drainage in a number of general surgery procedures such as superficial and total parotidectomy; thyroidectomy; tonsillectomy; pectoralis major myocutaneous flap dissection; axillary dissection; and lymphadenectomy have been reported with the use of Harmonic™.

The Harmonic™ has also been used in parotidectomy and maxillofacial surgery, but its use has been seldom mentioned in the field of plastic and reconstructive surgery. Recent use of the Harmonic™ has shown promise in plastic and reconstructive surgery in dissection of the pectoralis major myocutaneous flap and total body lifts.

Comparisons: The Harmonic™ vs. Electro Surgery in Lower Body Lift procedures.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for this clinical research study must fulfill all of the following criteria:

* Elect to undergo a Lower Body Lift procedure for post-obesity reasons;
* Able to comprehend and sign the study informed consent form;
* Able to return for all study mandated visits;
* Be a male or female greater than or equal to 18 years of age;
* Obtain medical clearance for a Lower Body Lift procedure according to institutional requirements.

Exclusion Criteria:

Subjects with any of the following criteria are not eligible to participate in this clinical research study:

* American Society Anesthesiologists (ASA) Classification of Physical Status greater than III;
* Current smoker (documented abstinence of 3 months);
* Documented current use of steroids or anti-inflammatory medications (within the past month) and no history of prolonged usage (for 1 month in the past 3 months);
* Diabetes mellitus (requiring treatment within the past year);
* Need of concomitant surgical procedures in which the wound drainage would interconnect with the wound regions studied by the trial (with the exception of liposuction);
* Presence of ventral or umbilical hernia requiring repair with the use of prosthetic material (e.g. mesh);
* Morbid obesity (Body Mass Index ≥ 40);
* At risk for ischemia due to presence of obstruction of the arterial blood supply or inadequate blood flow;
* Presence of scars that could limit flap advancement or that could not be completely excised;
* Current diagnosis or history of any disease that would impair the healing process;
* Current diagnosis or history of immune system disorders;
* Documented history of bleeding disorders;
* Presence of uncontrolled hypertension;
* Pregnant or lactating;
* Being treated with anticoagulants including aspirin within 7 days prior to surgery (a washout period of 7 days will be required); or
* Participation in any other clinical studies within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post massive weight loss
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al Aly, MD, Principal Investigator — Iowa City Plastic Surgery; Dirk Richter, MD, Principal Investigator — Facharzt für Plastische Chirurgie
Locations (2):
- Dr. Al Aly, Coralville, Iowa, United States
- Abteilung für Plastische und Ästhetische Chirurgie, Wesseling, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Harmonic® Technology: Harmonic® Sharp Curved Blade (HF105) instruments are indicated for soft tissue incisions when bleeding control and minimal thermal injury are desired. The instrument can be used as an adjunct to or substitute for electrosurgery, lasers, and steel scalpels in general, plastic, gynecologic, exposure to orthopedic structures (such as spine and joint space) and thoracic surgery.
  The Harmonic® Synergy™ Curved Blade (SNGCB) instruments are indicated for soft tissue incisions when bleeding control and minimal thermal injury are desired. The instruments can be used as an adjunct to or substitute for electrosurgery, lasers, and steel scalpels in general, plastic, gynecologic, exposure to orthopedic structures, Ear Nose and Throat (ENT), including tissues of the soft palate, oral structures, and oropharyngeal airway, and thoracic surgery, including mobilization of the Internal Mammary Artery.
  These devices were not modified from their commercially available specifications.
Period: Overall Study
Arm/Group | Electro Surgery | Harmonic® Technology
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electro Surgery | Harmonic® Technology | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.13 (10.239) | 38.13 (8.105) | 38.63 (9.088)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
  Germany | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Total Volume (mL) From the Time of Drain Placement to Time of Drain Removal
Description: Postoperative serous drainage volume was measured in milliliters and defined as the volume of serous fluid collected from the wound drains installed after the study procedure
Time Frame: From the time of drain placement to time of drain removal (</= 770 hours)
Population: ITT
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Electro Surgery | Harmonic® Technology
Number analyzed (Participants) | 15 | 15
milliliter | 2163.03 (756.295) | 1863.60 (1471.390)

2. Secondary Outcome: Total Number of Hours From Drain Placement to Drain Removal
Description: Total number of hours from drain placement to drain removal
Time Frame: From drain placement to drain removal (</= 770 hours)
Population: terminated study
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Electro Surgery | Harmonic® Technology
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Electro Surgery | Harmonic® Technology
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15
Other Adverse Events (participants affected / at risk) | 14/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electro Surgery (N=15) | Harmonic® Technology (N=15)
dyspnoea, MedDRA Version 10.0 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
wound dehiscence, MedDRA 10.0 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electro Surgery (N=15) | Harmonic® Technology (N=15)
ANAEMIA ,MedDRA 10.0 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vertigo, MedDRA 10.0 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Nausea; MedDRA 10.0 (Gastrointestinal disorders) | 6 (6) | 6 (6)
constipations; MedDRA 10.0 (Gastrointestinal disorders) | 2 (2) | 2 (2)
Chills; MedDRA 10.0 (General disorders) | 1 (1) | 1 (1)
impaired healing; MedDRA 10.0 (General disorders) | 1 (1) | 1 (1)
Pyrexia; MedDRA 10.0 (General disorders) | 1 (1) | 1 (1)
Application site reaction; MedDRA 10.0 (General disorders) | 0 (0) | 1 (1)
Application site vesicles; MedDRA 10.0 (General disorders) | 0 (0) | 1 (1)
fatigue; MedDRA 10.0 (General disorders) | 0 (0) | 1 (1)
sinusitis;MedDRA 10.0 (Infections and infestations) | 0 (0) | 1 (1)
infection; MedDRA 10.0 (Infections and infestations) | 1 (1) | 0 (0)
staphyloccal infection; MedDRA 10.0 (Infections and infestations) | 1 (1) | 0 (0)
vaginal infection; MedDRA 10.0 (Infections and infestations) | 0 (0) | 1 (1)
abdominal distension; MedDRA 10.0 (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal haematoma; MedDRA 10.0 (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal rigidity; MedDRA 10.0 (Gastrointestinal disorders) | 1 (1) | 0 (0)
seroma; MedDRA 10.0 (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
anaemia postoperative; MedDRA 10.0 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
device leakage; MedDRA 10.0 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
medical device pain; MedDRA 10.0 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome; MedDRA 10.0 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
procedural nausea; MedDRA 10.0 (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
body temperature increased; MedDRA 10.0 (Investigations) | 1 (1) | 1 (1)
blood pressure decreased; MedDRA 10.0 (Investigations) | 0 (0) | 1 (1)
lumbar puncture; MedDRA 10.0 (Investigations) | 1 (1) | 0 (0)
fluid retention; MedDRA 10.0 (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
pain in extremity; MedDRA 10.0 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dizziness; MedDRA 10.0 (Nervous system disorders) | 1 (1) | 5 (5)
headache; MedDRA 10.0 (Nervous system disorders) | 0 (0) | 1 (1)
hypoaesthesia; MedDRA 10.0 (Nervous system disorders) | 1 (1) | 0 (0)
intercranial hypotension; MedDRA 10.0 (Nervous system disorders) | 1 (1) | 0 (0)
syncope; MedDRA 10.0 (Nervous system disorders) | 0 (0) | 1 (1)
anxiety; MedDRA 10.0 (Psychiatric disorders) | 1 (1) | 1 (1)
insomnia; MedDRA 10.0 (Psychiatric disorders) | 0 (0) | 1 (1)
urge incontinence; MedDRA 10.0 (Renal and urinary disorders) | 1 (1) | 0 (0)
perineal pain; MedDRA 10.0 (Reproductive system and breast disorders) | 1 (1) | 0 (0)
nasal congestion; MedDRA 10.0 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
respiratory disorder; MedDRA 10.0 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pruritis; MedDRA 10.0 (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6)
blister; MedDRA 10.0 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
erythema; MedDRA 10.0 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
hypertension; MedDRA 10.0 (Vascular disorders) | 0 (0) | 1 (1)
ischaemia; MedDRA 10.0 (Vascular disorders) | 0 (0) | 1 (1)
thrombosis; MedDRA 10.0 (Vascular disorders) | 0 (0) | 1 (1)
Application site Excoriation, medDRA 10.0 (General disorders) | 1 (1) | 0 (0)
Asthenia, MedDRA 10.0 (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has at least 60 days for review to ensure non disclosure of Confidential information. If Study is a multicenter study, PI agrees that the first publication shall include results from all PIs contributing data. If multicenter publication is not submitted within 12 months,or after Sponsor confirms there will be no multicenter Study publication, the Institution and/or such PI may publish the results from their respective site individually in accordance with this paragraph.